CLINICAL TRIAL: NCT03929055
Title: Efficacy of High Velocity Nasal Insufflation Compared With Venturi Mask and Helmet CPAP in Acute Respiratory Failure
Brief Title: Efficacy of High Velocity Nasal Insufflation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Davide Chiumello, Prof, University of Milan
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HFNC
Record Dates: First submitted 2019-04-20; First posted 2019-04-26 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Acute Respiratory Failure; Diaphragmatic Function; Esophageal Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- venturi mask (Active Comparator): oxygen is delivered by venturi mask to achieve peripheral oxygen saturation of al least 92%
  Interventions: Device: Physiological assesment
- HFNC (Active Comparator): HFNC is set to obtain the same oxygen fraction of venturi mask and flow of 40l/min
  Interventions: Device: Physiological assesment
- CPAP (Active Comparator): Helmet CPAP is set to obtain the same esophageal pressure variation during HFNC step
  Interventions: Device: Physiological assesment

INTERVENTIONS:
Device: Physiological assesment — 1. Arterial blood gas analysis.
  2. esophageal pressure variation during inspiration and expiration
  3. Arterial blood pressure, central venous pressure (CVP), heart rate.
  4. diaphragmatic contraction detected by ultrasound

SUMMARY:
The purpose of this study is to assess the effect of HFNC on esophageal pressure and diaphragmatic function in patients with acute respiratory failure

DETAILED DESCRIPTION:
In recent years, new devices that deliver totally conditioned gas through a nasal cannula at high flow have emerged as a safe and useful supportive therapy in many clinical situations. High flow nasal cannula (HFNC) supportive therapy is one such technique that exerts its potential benefits through a variety of mechanisms. In the last two decades, HFNC supportive therapy has emerged as a safe, useful therapy in patients with respiratory failure. Several mechanisms are known to contribute to oxygenation improvement and carbon dioxide reduction, which are the main potential benefits of using HFNC therapy. However, the exact contributions of each mechanism have not been conclusively established and these may, in fact, vary from one patient to another. Recently several clinical trials have analyzed the effectiveness of HFNC therapy in different clinical situations and have reported promising results such as the potential to improve clinical outcomes. However, the physiologic mechanisms underlying the clinical benefits of HFNC are still poorly understood in adult patients. Basic clinical monitoring during HFNC therapy demonstrated rapid improvement of oxygenation and reduction of dyspnea in comparison to a standard facial mask. Findings in other populations indicate that advanced respiratory monitoring might demonstrate other specific physiologic effects such as the reduction in inspiratory effort and increment in lung volume that may prevent respiratory muscle exhaustion and lower the tidal volume/end expiratory lung volume (EELV) ratio. Moreover, It has been hypothesized that the continuous administration of a very high flow of gas flushes the carbon dioxide (CO2) out of the upper respiratory airway, avoiding the re-inhalation of the previous exhaled gas. A randomized, crossover, experimental study with neonatal piglets with lung injury treated with continuous positive airway pressure (CPAP; minimal leak) or a HFNC with a high or low degree of leak around the nasal prongs showed that under both HFNC leak conditions PaCO2 decreased and oxygen arterial pressure (PaO2) increased with increasing flow. This effect of nasopharyngeal dead space washout was associated more with increases in flow rates than with increases in pressure. Thus, compared with the masks used with conventional oxygen delivery devices, nasal prongs reduce dead space.

Additionally, high velocity flows likely reduce inspiratory resistance and allow the patient to breathe from their dead space, rather than through it. This is how high velocity Nasal Insufflation helps reduce work of breathing, respiratory rate and assists in increasing alveolar ventilation efficiency.

The relative contribution of the patient's effort during assisted breathing is difficult to measure in clinical conditions, and the diaphragm, the major muscle of inspiratory function, is inaccessible to direct clinical assessment. Several methods have been used in the research setting to assess diaphragmatic contractile activity. Bedside ultrasonography, which is already crucial in several aspects of critically illness, has been recently proposed as a simple, non-invasive method of quantification of diaphragmatic contractile activity . Ultrasound can be used to determine diaphragm excursion which may help to identify patients with diaphragm dysfunction Ultrasonographic examination can also allow for the direct visualization of the diaphragm thickness in its zone of apposition. Thickening during active breathing has been proposed to reflect the magnitude of diaphragmatic effort, similarly to an ejection fraction of the heart. In spontaneously breathing patients, thickness fraction was shown to be positively related to tidal volume and thickness measurements during spontaneous breathing may be influenced by lung volume in a non-linear relationship, and diaphragmatic thickening was shown to be more pronounced above 50% of vital capacity. It seems reasonable to expect that the high flow nasal cannula may modify the thickness or diaphragm thickening and its excursion depend on the level of positive end expiration pressure generated. On the other hand, it could also happen that with a relevant increase in tidal volume the diaphragmatic excursion may remain constant. The most likely explanation is that a higher portion of the tidal volume (VT) is distributed to the non-dependent lung region due to better compliance of this area, as recently shown with electrical impedance tomography analysis. Another possible explanation is that patients' respiratory muscles could be over-assisted and the diaphragm may be passively displaced downward by simply improving gas exchange efficacy.

The aim of the present study is to compare the HFNC, Helmet continues positive airway pressure (CPAP) and venturi mask on the inspiratory effort, respiratory rate, gas exchange, level of dyspnea and diaphragmatic function evaluated by US in a group of patients with acute respiratory failure (ARF).

Inclusion and exclusion criteria The study has been submitted to our local ethics committee and patients will receive their written informed consent. All consecutive patients with acute respiratory failure presenting as respiratory rate higher than 25-30; Pao2 / oxygen inspiratory fraction (FiO2) ratio less than 300 supported with venturi mask at 30% Fio2. Patients will be exclude if there will be present one of the following conditions: PaO2/FiO2 less than 100; hemodynamic instability (mean arterial pressure lower than 60 mmHg after fluid challenge) and impossibility to insert the esophageal monitoring. Sample size calculation is based on the results of the study by Mauri, in which the application of HFNC at a similar flow rate to patients suffering from acute hypoxemic respiratory failure determined a reduction in esophageal pressure swing from 9.4+-4.1 to 7.9+-3.0. If the investigators hypothesize that a similar effect size is present in our patient population, a sample size of 25 patients will be necessary to achieve a level of significance of 0.05, with a 0.8 power, for a repeated-measures study design. Normally distributed variables are expressed as mean ± standard deviations and were analysed by a paired t-test. Non-normally distributed variables are expressed as medians and were compared by Wilcoxon's signed rank test. Correlations were analysed by Pearson's coefficient. A level of p<0.05 (two-tailed) was considered statistically significant.

Experimental settings and Measurements A cross over study. Patients will enter in the three study phases with the same set clinical FiO2 for 20 minutes: standard Venturi oxygen mask with FiO2 regulated to achieve 90-04% of oxygen saturation (SpO2) with a flow rate of 35-40 Litters/minute (L/m); high velocity nasal insufflation (Precision Flow) with optimized gas flow; Helmet CPAP with positive end expiatory pressure (PEEP) set to reach the same esophageal swing obtained with HFNC. Using a small-bore nasal cannula the study will start with a flow rate set to 35 L/min, with a starting temperature between 35°C and 37°C and FIO2 at 1.0. Adjustments in flow (within the range of 25 L/min to 40 L/min) and temperature (typically between 35°C to 37°C) are made to alleviate respiratory distress and optimize comfort; FIO2 was titrated to maintain SpO2 at 90-94%.

At enrolment, the investigators will collect the patients' main demographics and clinical data. An esophageal balloon catheter will be placed in the esophagus, as demonstrated by the appearance of cardiac artefacts and appropriate negative swings of pressure tracings during inspiration. Esophageal pressure waveforms will be continuously recorded by a dedicated data acquisition system throughout the study. At each steps ultrasonography of the diaphragm will be performed using an ultrasound machine (GE Healthcare) equipped with a high-resolution 10-megahertz (MHz) linear probe and a 7.5-MHz convex phased-array probe. Images will be recorded for subsequent computer- assisted quantitative analysis performed by a trained investigator. The convex probe will be placed below the right costal margin along the mid-clavicular line, so that the ultrasound beam are perpendicular to the posterior third of the corresponding hemi-diaphragm, as previously described. Patients will be scanned along the long axis of the intercostal spaces, with the liver serving as an acoustic window. M-mode will then be used to display diaphragm excursion. Diaphragm thickness (DT) will be assessed in the zone of apposition of the diaphragm to the rib cage. The inferior border of the costophrenic sinus will be identified as the zone of transition from the artifactual representation of normal lung to the visualization of the diaphragm and liver. In this area, the diaphragm is observed as a three-layered structure: a non-echogenic central layer bordered by two echogenic layers, the peritoneum and the diaphragmatic pleurae.

ELIGIBILITY:
Inclusion Criteria:

* patient with acute respiratory failure, not intubated, who require non invasive mechanical ventilation

Exclusion Criteria:

* patients in which it is not possible to place the esophageal catheter or it is not possible to detect the diaphragm by ultrasound or it is not possible to apply the nasal cannula device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
effects of HFNC on esophageal pressure variation | one day
  the esophageal pressure will be measure using an esophageal ballon catheter. A decrease in esophageal pressure variation during HFNC treatment compared with CPAP

SECONDARY OUTCOMES:
effect of HFNC on diaphragmatic function | one day
  the diaphragmatic function will be detected using the ultrasound. An improvement in diaphragmatic contractility function as detected by the increase in its thickness ratio is expected during HFNC treatment compared with CPAP

CONTACTS AND LOCATIONS:
Locations (1):
- ASST-Santi Paolo e Carlo, San Paolo Hospital, Milan, Italy